CLINICAL TRIAL: NCT02804529
Title: A Comparison of Three Different Puncture Points to Establish the Pneumoperitoneum in Laparoscopic Gastrointestinal Surgery: A Randomized Prospective Trial
Brief Title: A Comparison of Three Different Entry Points to Establish the Pneumoperitoneum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Fanqiang Meng, MD. PhD., China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChinaJapanFH Meng001
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Laparoscopic Entry Technique
Keywords: Laparoscopic entry; Meng's point; Veress needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Meng's Point entry (Experimental): Meng's entry involved a 0.2 cm horizontal or vertical incision using the Veress needle in the cross of lateral border of the left rectus abdominis and rib arch.
  Interventions: Device: Veress needle
- Palmer's Point entry (Experimental): Palmer's entry involved a 0.2 cm horizontal or vertical incision with the Veress needle in the left midclavicular line approximately 3 cm caudal to the 10th rib
  Interventions: Device: Veress needle
- Periumbilllicus entry (Experimental): Periumbilllicus entry involved a 0.2 cm horizontal or vertical midline incision using the Veress needle in the lower or uper border of the umbilicus.
  Interventions: Device: Veress needle

INTERVENTIONS:
Device: Veress needle

SUMMARY:
The Palmer's point and periumbilical region are the common laparoscopic entry site to establish the pneumoperitoneum. In the present study, the investigators assess the safety and feasibility of Meng's point as a new laparoscopic entry site in cases to perform the gastrointestinal surgery.

This prospective and randomized study will compare the three entry techniques with regard to:

* Complications related to the entry technique
* Time taken to enter the abdomen.
* The number of attempts taken to enter the abdomen

DETAILED DESCRIPTION:
Patients of China-Japan Friendship Hospital that are having a laparoscopic surgery for general surgery purposes will participate in the study. Patients with previous abdominal surgeries will be excluded from the study. A patient information sheet will be provided and written consent will be obtained. Patients who give written consent will be randomized into the three arms of the trial. All patient information will be confidential and only be available to researches involved in the study. Only one attending surgeon of the General Surgery Department of China-Japan Friendship Hospital will participate in the study. 90 patients will be recruited over one year period and the data will be analysed by a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Any patient suitable for laparoscopic abdominal surgery

Exclusion Criteria:

* previous abdominal surgeries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Complications during entry in laparoscopy | During surgery

SECONDARY OUTCOMES:
Time to enter in the abdominal cavity | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fanqiang Meng, MD,CSCRS, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Granata M, Tsimpanakos I, Moeity F, Magos A. Are we underutilizing Palmer's point entry in gynecologic laparoscopy? Fertil Steril. 2010 Dec;94(7):2716-9. doi: 10.1016/j.fertnstert.2010.03.055. Epub 2010 May 10. PMID 20452584
- [Background] Angioli R, Terranova C, De Cicco Nardone C, Cafa EV, Damiani P, Portuesi R, Muzii L, Plotti F, Zullo MA, Panici PB. A comparison of three different entry techniques in gynecological laparoscopic surgery: a randomized prospective trial. Eur J Obstet Gynecol Reprod Biol. 2013 Dec;171(2):339-42. doi: 10.1016/j.ejogrb.2013.09.012. Epub 2013 Sep 23. PMID 24103531
- [Background] Ahmad G, Gent D, Henderson D, O'Flynn H, Phillips K, Watson A. Laparoscopic entry techniques. Cochrane Database Syst Rev. 2015 Aug 31;8:CD006583. doi: 10.1002/14651858.CD006583.pub4. PMID 26329306